CLINICAL TRIAL: NCT00170378
Title: The Use of Low Molecular Weight Heparin in Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSR #02-2113
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2012-10

CONDITIONS: Brain Injury; Venous Thrombosis
Keywords: Enoxaparin; Safety
MeSH Terms: conditions — Brain Injuries; Venous Thrombosis | interventions — Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
To study the safety and efficacy of early administration of Low Molecular Weight Heparin to patients with traumatic brain injury.

DETAILED DESCRIPTION:
Venous thromboembolic (VTE) prophylaxis in trauma patients is a critical clinical problem. Patients with traumatic brain injury usually have effective VTE prophylaxis withheld secondary to concerns of exacerbating intracranial hemorrhage. This study examines the safety and efficacy of early administration (within 24 hrs of admission) of low molecular weight heparin to this patient population with very high VTE risk.

ELIGIBILITY:
Inclusion Criteria:

* Blunt traumatic brain injury (Marshall II-V)
* Stable 6 hr. head CT
* Stable hemoglobin

Exclusion Criteria:

* Premorbid coagulopathy
* Pregnancy
* < 18 y.o.
* Need for therapeutic anticoagulation
* Heparin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-12; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Safety: Assess if early administration of LMWH exacerbates intracranial hemorrhage.

SECONDARY OUTCOMES:
Efficacy: Demonstrate effectiveness of dosing regimen in preventing VTE.

CONTACTS AND LOCATIONS:
Overall Officials: John K. Cumming, M.D., Principal Investigator — Hennepin County Medical Center/MinneapolisMRF
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, Gearhart MM, Zurick A, Zuccarello M, James L, Luchette FA. Preliminary report on the safety of heparin for deep venous thrombosis prophylaxis after severe head injury. J Trauma. 2002 Jul;53(1):38-42; discussion 43. doi: 10.1097/00005373-200207000-00008. PMID 12131387
- [Background] Norwood SH, McAuley CE, Berne JD, Vallina VL, Kerns DB, Grahm TW, Short K, McLarty JW. Prospective evaluation of the safety of enoxaparin prophylaxis for venous thromboembolism in patients with intracranial hemorrhagic injuries. Arch Surg. 2002 Jun;137(6):696-701; discussion 701-2. doi: 10.1001/archsurg.137.6.696. PMID 12049541
- [Background] Norwood SH, McAuley CE, Berne JD, Vallina VL, Kerns DB, Grahm TW, McLarty JW. A potentially expanded role for enoxaparin in preventing venous thromboembolism in high risk blunt trauma patients. J Am Coll Surg. 2001 Feb;192(2):161-7. doi: 10.1016/s1072-7515(00)00802-4. PMID 11220715